CLINICAL TRIAL: NCT00935909
Title: Use of Vein Viewer for Insertion of Peripheral Venous Cannula in Pediatric Patients With Difficult Intravenous Access.
Status: Completed | Type: Observational
Sponsor: Peter Szmuk (Other)
Collaborators: Luminex Corporation (Industry); Outcomes Research Consortium (Other)
Responsible Party: Sponsor-Investigator, Peter Szmuk, Professor, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Other Study IDs: 112008-014
Record Dates: First submitted 2009-07-02; First posted 2009-07-09 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: IV Cannulation
Keywords: IV cannulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary purpose of this prospective, randomized trial is successful intravenous (IV) cannulation on first attempt with the use of either the Vein Viewer (VV) or standard cannulation method. The secondary purpose is to find out if there is a difference in the total time to successful cannulation.

DETAILED DESCRIPTION:
A single initial data page will be filled out by one of the study team members present with the IV Team at the time of the cannulation. The data from these forms will be entered by the investigator or research assistant into a database maintained only for this study. There will be two groups in this randomized study. One group will receive IV cannulation with the VV and the second group will receive standard cannulation without the VV. The chance of receiving either treatment is based on randomly generated computer codes, unknown by the IV team. We want to evaluate successful IV cannulation on first attempt as well as the time taken for cannulation. All documents will be de-identified of data that contains HIPAA protected health information (PHI) at the end of the study. We estimate approximate enrollment to be 790 children. The study is expected to last 12 months and will only be conducted at Children's Medical Center Dallas.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 0-18 requiring IV cannula (ASA 1-4) with a modified DIVA score ≥ 2 at the time of assessment

Exclusion Criteria:

* Patients with visible veins will be excluded from the study as well as patients with known difficult IV access which are scheduled for PICC line placement.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The floor patients meeting the inclusion/exclusion criteria that need an IV
Sampling Method: Probability Sample
Enrollment: 603 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Successful IV cannulation on the first attempt | Time of cannulation will be measured from the application of the tourniquet until successful IV cannulation.

SECONDARY OUTCOMES:
Total time to successful IV cannulation | Time of cannulation will be measured from the application of the tourniquet until successful IV cannulation.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Szmuk, MD, Principal Investigator — UT Southwestern
Locations (1):
- Children's Medical Center Dallas, Dallas, Texas, United States